CLINICAL TRIAL: NCT06600854
Title: Clinical Feasibility of BoneTape: a Novel Approach for Zygomaticomaxillary Fracture Fixation
Brief Title: BoneTape Feasibility Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cohesys Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-CMF-001
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Zygomaticomaxillary Complex Fracture; Zygomatic Fractures; Zygoma Fracture
Keywords: Craniomaxillofacial; Zygomaticomaxillary; Fracture; Medical Device; Fracture Fixation; Zygomatic Fractures; Implant; BoneTape™
MeSH Terms: conditions — Zygomatic Fractures; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BoneTape (Experimental)
  Interventions: Device: BoneTape

INTERVENTIONS:
Device: BoneTape — BoneTape is a craniofacial fracture repair device intended for use in the fixation of non-load-bearing bones of the craniofacial and midfacial skeleton. It can be used in skeletally mature individuals but is not intended for use in the mandible and/or full load bearing procedures. It is composed of: 1) BoneTape implant ("device"), and 2) BoneTape applicator ("applicator").

SUMMARY:
This study aims to evaluate the safety, effectiveness, and usability of BoneTape, an innovative medical device designed to fix facial bone fractures, specifically in the zygomaticomaxillary (midface) region. Zygomaticomaxillary fractures, often caused by trauma like car accidents or falls, require surgery to align and stabilize the bones for proper healing. Traditional methods use metal plates and screws, which can be complicated to install, over-engineered for the area, and may lead to complications, requiring additional surgeries.

BoneTape is a new, resorbable (biodegradable) device that offers a simpler, potentially safer alternative. Unlike traditional metal hardware, BoneTape is a flexible, thin plate that can be easily cut to the required shape during surgery and applied directly to the bone using a special tool that anchors it without needing to drill or screw holes. This process significantly simplifies the surgical procedure, reduces the time needed for fixation, and avoids complications associated with drilling into healthy bone tissue.

Study Objectives:

Feasibility: Determine if BoneTape can be successfully used to stabilize midfacial fractures.

Effectiveness: Assess the ability of BoneTape to help bones heal properly without additional complications.

Safety: Monitor and evaluate any adverse events related to the use of BoneTape.

Study Design:

The study is designed as a single-arm, cohort study.

Participants will undergo baseline pre-operative assessments, including clinical exams, CT scans, and pain questionnaires. BoneTape will be applied during surgery, and post-operative assessments will take place within 24 hours. Follow-up visits will occur at 1 week, 6 weeks, 24 weeks, and 12 months to monitor the healing process, assess pain levels, and check for any adverse events.

Eligibility Criteria:

Inclusion:

Adults with a unilateral, non-comminuted (not broken into multiple pieces) zygomaticomaxillary fracture requiring surgery.

Must be skeletally mature, able and willing to attend follow-up visits, and provide informed consent.

Exclusion:

Patients with critically sized bone defects, fractures requiring orbital floor surgery, pregnancy, certain medical conditions impairing bone healing, or those unwilling or unable to follow the study procedures.

Study Duration:

The total study duration is expected to be 21-24 months, including the 12-month follow-up period for each participant.

Outcome Measures:

The primary outcomes include the feasibility of the procedure (successful use of BoneTape without additional hardware), early effectiveness (bone healing and stability at 6 and 24 weeks), and safety (rate and type of adverse events up to 24 weeks). Secondary outcomes will assess long-term safety and effectiveness at 12 months, patient-reported outcomes on pain, and physician feedback on device usability.

This study is a critical step in evaluating BoneTape as a potential alternative to current facial bone fixation methods, potentially improving surgical outcomes and patient quality of life by reducing the complexity of procedures and minimizing the need for additional surgeries.

ELIGIBILITY:
Inclusion Criteria: Patients who meet all of the following criteria will be eligible for inclusion in the study:

* Have a non-comminuted unilateral unstable zygomatico-maxillary fracture at one or more sites requiring operative intervention;
* Are skeletally mature;
* Able and willing to return for follow-up visits;
* Able and willing to provide informed assent or consent.

Exclusion Criteria: Patients who meet any of the following criteria will be excluded from the study:

* Present critically sized bone defects*, as determined by the investigator;
* Have a fracture of the orbital floor requiring operative intervention;
* Are pregnant;
* Are not willing or able to participate in follow-ups;
* In whom the general health and/or medication could impair bone healing, as determined by the investigator;
* Are pre-diagnosed with osteoporosis or are diagnosed by the investigator during baseline pre-operative assessment;
* Are smokers;
* Have a pacemaker;
* Have active or latent infection.

  * A critically sized bone defect refers to a bone injury or loss that is of sufficient size such that it exceeds the natural regenerative capacity of the bone, rendering spontaneous healing unlikely over the patient's lifetime. The determination of a 'critical size' is case-dependent and requires clinical judgment, taking into account factors such as the specific bone affected, its location, the blood supply to the area, the presence of surrounding soft tissues, and the patient's overall health status.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2027-01-05 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Intervention
  Procedure success in target population.
Early Efficacy | Intervention to 24-weeks post-op
  Clinical and radiographic bone union
Early Safety | Intervention to 24-weeks post-op
  Rate of adverse events

SECONDARY OUTCOMES:
Safety and Efficacy | Intervention to 12-months post-op
  Rate of adverse events and clinical examination
Pain | Baseline to 12 months post-op
  Pain scored using Numerical rating Scale
Physician usability and feedback | Intervention
  Surgeon will complete a specific questionnaire to rate and provide feedback

OTHER OUTCOMES:
Facial photographs | Baseline to 12 months post-op
Operative time | Intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No